CLINICAL TRIAL: NCT07189585
Title: Change in LPS With Inulin Supplementation and Its Association With Knee Pain Among Older Adults With Osteoarthritis
Brief Title: Inulin Supplementation for Reducing Inflammation and Knee Pain in Older Adults With Osteoarthritis
Acronym: OA-INULIN
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: VA Connecticut Healthcare System (U.S. Federal Agency); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Evelyn Hsieh Donroe, Associate Professor of Medicine, Yale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000040523; 174626 (Other: FDA IND); 1R61AT013472-01 (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2025-09-16; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Knee Osteoarthritis
Keywords: Inulin; Prebiotic; Lipopolysaccharide; Inflammation; Knee pain; Older adults
MeSH Terms: conditions — Osteoarthritis, Knee; Inflammation | interventions — Inulin; maltodextrin

STUDY DESIGN:
Intervention Model Description: Participants are randomized in a 1:1:1 ratio to placebo, 10 g/day inulin, or 15 g/day inulin for 8 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Inulin and placebo are identical in appearance, taste, and packaging. Randomization is managed by the investigational pharmacy; study staff, investigators, and participants remain blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Maltodextrin) (Placebo Comparator): Participants receive maltodextrin powder in identical sachets. Dose is escalated over 2 weeks to match the dosing schedule of the inulin arms (5 g daily for 3 days, 10 g daily for 4 days, then 15 g daily). Sachets are mixed with food or beverage and taken once daily with the largest meal, for 8 weeks.
  Interventions: Drug: Maltodextrin (Placebo)
- Inulin 10 g/day (Experimental): Participants receive inulin powder in identical sachets. Dose is escalated to 10 g daily (5 g daily for 3 days, then 10 g daily for 4 days). After Week 2, participants continue with one 15 g sachet containing a 2:1 blend of inulin and maltodextrin, providing a daily dose of 10 g inulin. Sachets are mixed with food or beverage and taken once daily with the largest meal, for 8 weeks.
  Interventions: Drug: inulin
- Inulin 15 g/day (Experimental): Participants receive inulin powder in identical sachets. Dose is escalated to 15 g daily (5 g daily for 3 days, 10 g daily for 4 days, then 15 g daily). Sachets are mixed with food or beverage and taken once daily with the largest meal, for 8 weeks.
  Interventions: Drug: inulin

INTERVENTIONS:
Drug: inulin — Inulin is a fermentable prebiotic fiber derived from chicory root. For this study, inulin is packaged into single-dose sachets containing 5 g, 10 g, or 15 g of powder. Participants in the 10 g arm escalate from 5 g/day for 3 days to 10 g/day, then continue with sachets containing a 2:1 blend of inulin and maltodextrin to provide a daily 10 g inulin dose. Participants in the 15 g arm escalate from 5 g/day for 3 days, 10 g/day for 4 days, then 15 g/day for the remaining 8 weeks. Sachets are mixed with food or beverage and taken once daily with the largest meal.
  Other Names: Orafti® Inulin; BENEO-Orafti
  Arms: Inulin 10 g/day; Inulin 15 g/day
Drug: Maltodextrin (Placebo) — Maltodextrin is a carbohydrate powder widely used as a food additive. For this study, maltodextrin is used as the placebo comparator. It is packaged into single-dose sachets identical in appearance and taste to inulin sachets. Participants receive escalating doses (5 g/day for 3 days, 10 g/day for 4 days, then 15 g/day) for a total of 8 weeks. Sachets are mixed with food or beverage and taken once daily with the largest meal.
  Other Names: Placebo
  Arms: Placebo (Maltodextrin)

SUMMARY:
This study will test whether inulin, a type of dietary fiber, can reduce inflammation in older adults with knee osteoarthritis. Inflammation in the body may contribute to both joint pain and the progression of osteoarthritis. Inulin is a prebiotic fiber that may improve gut health and reduce lipopolysaccharide (LPS), a marker of bacterial products in the blood that is linked to inflammation.

In this trial, participants with knee osteoarthritis will be randomly assigned to receive either inulin or a placebo (maltodextrin) for 8 weeks. The study will measure changes in blood LPS levels, knee pain, and other markers of inflammation. The goal is to determine whether inulin supplementation can improve pain and reduce inflammation in people with knee osteoarthritis.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a leading cause of pain and disability among older adults. Low-grade systemic inflammation has been implicated in OA pathogenesis, and bacterial products such as lipopolysaccharide (LPS) translocated from the gut microbiome may contribute to joint inflammation. Inulin-type fructans are non-digestible carbohydrates classified as prebiotic fibers. By modulating the gut microbiome, inulin has been shown to promote the growth of beneficial bacteria and to increase short-chain fatty acid (SCFA) production, which may help reduce systemic LPS levels and inflammation.

This is a single-center, randomized, double-blind, placebo-controlled clinical trial of participants aged 40 years or older with radiographically confirmed knee OA and significant knee pain. Participants will be randomized in a 1:1:1 ratio to receive 10 g/day inulin, 15 g/day inulin, or placebo (maltodextrin) for 8 weeks. The primary outcome is change in serum LPS from baseline to 8 weeks in the combined inulin groups compared to placebo.

The study hypothesis is that inulin supplementation will reduce circulating LPS and improve knee pain outcomes, supporting the role of gut microbiome modulation in the management of OA-related inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Stated willingness to comply with all study procedures and availability for the duration of the study (8 weeks).
* Male or female, aged ≥ 40 years.
* Established patient in the VA Connecticut Healthcare System
* At least one knee with pain severity in the past week ≥ 4/10 on numerical rating scale (NRS)
* Self-reported knee pain on most days of the prior month.
* Diagnosed with knee osteoarthritis (Kellgren-Lawrence grade 2-4 on radiographic imaging within the past 2 years).
* Ability to take oral powder supplements and willingness to adhere to the inulin/placebo daily regimen.
* Agreement to adhere to lifestyle considerations (see Section 5.3) throughout study duration, including maintenance of current diet, physical activity, and avoidance of new dietary supplements or complementary therapies.
* English-speaking and able to provide informed consent.
* For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to continue such method during study participation.

Exclusion Criteria:

* Current diagnosis of pre-diabetes (impaired glucose tolerance) or diabetes mellitus (Type 1 or Type 2).
* Use of antibiotics within the past 6 months.
* Current use of medications known to significantly impact the gut microbiome (e.g., proton pump inhibitors, disease-modifying antirheumatic drugs, GLP-1 receptor agonists).
* Use of anti-inflammatory dietary supplements (e.g., turmeric, omega-3 fatty acids) within the past 30 days.
* Participation in another interventional study or use of an investigational drug within the past 30 days.
* Current use of complementary or integrative therapies for knee OA including tai chi, acupuncture or yoga.
* Known allergy or intolerance to components of the study intervention, including inulin or maltodextrin.
* The presence of significant gastrointestinal disease that may interfere with the intervention or outcomes, such as inflammatory bowel disease or active peptic ulcer disease.
* Any medical, psychological, or behavioral condition that, in the opinion of the investigators, would place the participant at undue risk, interfere with study participation or adherence, or compromise data integrity.
* Current diagnosis of alcohol use disorder
* Pregnancy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in serum lipopolysaccharide (LPS) concentration from baseline to 8 weeks | Baseline and 8 weeks
  Serum LPS levels will be measured at baseline and at 8 weeks to evaluate the effect of inulin supplementation compared to placebo.

SECONDARY OUTCOMES:
Change in serum LPS concentration between 10 g and 15 g inulin groups | Baseline and 8 weeks
  Dose-response effect of inulin supplementation on serum LPS levels.
Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Baseline and 8 weeks
  Self-reported knee pain and function will be measured using the WOMAC scale. Higher scores indicate worse pain, stiffness, and functional limitations. Total possible score of 0-96.

OTHER OUTCOMES:
Change in systemic inflammatory biomarkers | Baseline and 8 weeks
  Changes in circulating CRP, IL-6, TNF-α, and LBP concentrations will be measured.
Change in synovial fluid LPS concentration | Baseline and 8 weeks
  Synovial fluid will be collected at baseline and 8 weeks to assess changes in LPS levels.
Change in knee pain | Baseline and 8 weeks
  Knee pain will be assessed using the Numeric Rating Scale (NRS). Total score range 0-10 with higher scores indicating more severe pain.
Adherence rate (% sachets taken) | Baseline through Week 8
  Adherence to the assigned intervention will be assessed by calculating the percentage of study sachets taken during the 8-week intervention period. Participants will be asked to return unused sachets at each visit. Adherence will be expressed as the number of sachets consumed divided by the total number expected.

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn Hsieh, MD, PhD, Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, West Haven Campus, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study is conducted within the Veterans Affaire system, which prohibits release of participant-level data outside of the VA firewall. However, de-identified aggregate group-level data, study protocol, data collection instruments, and analytic code will be made available to qualified researchers upon request in accordance with NIH Data Management and Sharing policy.